CLINICAL TRIAL: NCT00048555
Title: A Phase I/II Trial of IDEC-114 (Anti-CD80 Monoclonal Antibody) in Combination With Rituxan® for Patients With Relapsed or Refractory, Follicular Lymphoma
Brief Title: Safety and Efficacy of IDEC-114 in Combination With Rituxan in the Treatment of Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Study MD, Biogen Idec
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114-21; NCT00056043 (obsolete NCT alias)
Record Dates: First submitted 2002-11-01; First posted 2002-11-05 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-01

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — galiximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: IDEC-114

INTERVENTIONS:
Drug: IDEC-114 — Dose Group 1 - 125 mg/m2 x 4 infusions & 375 mg/m2 Rituxan x 4 infusions Dose Group 2 - 250 mg/m2 x 4 infusions & 375 mg/m2 Rituxan x 4 infusions Dose Group 3 - 375 mg/m2 x 4 infusions & 375 mg/m2 Rituxan x 4 infusions Dose Group 4 - 500 mg/m2 x 4 infusions & 375 mg/m2 Rituxan x 4 infusions

SUMMARY:
To determine what side effects and what clinical effect, if any, the administration of this investigational product, IDEC-114 in combination with Rituxan® [Rituxan® as a single agent is approved by the United States Food and Drug Administration (FDA) to treat patients with relapsed or refractory follicular NHL], has in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Signed IRB-approved informed consent
* Greater than or equal to 18 years of age
* Proof of follicular lymphoma
* Progressive disease requiring treatment after at least 1 prior standard therapy
* Acceptable hematologic status, liver function, and renal function
* Patients of reproductive potential must agree to follow accepted birth control methods during treatment and for 3 months after completion of treatment

Exclusion Criteria:

* No response to prior Rituxan® or Rituxan®-containing regimen
* Presence of CLL or CNS lymphoma
* Known history of HIV infection or AIDS
* Prior diagnosis of aggressive NHL or mantle-cell lymphoma
* Serious nonmalignant disease
* Pregnant or currently breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2002-11; Primary Completion 2004-03 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To characterize the safety profile and to define the dose of galiximab to be used for the Phase II portion of the study | March 2010

SECONDARY OUTCOMES:
To evaluate PK | March 2010
To evaluate efficacy | March 2010
To monitor for the presence of human anti galiximab antibody and human antichimeric antibody formation | March 2010

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Research site, Birmingham, Alabama
  - Research site, Tucson, Arizona
  - Research site, Los Angeles, California
  - Research site, Newport Beach, California
  - Research site, San Diego, California
  - Research site, Aurora, Colorado
  - Research site, Washington D.C., District of Columbia
  - Research site, Tampa Bay, Florida
  - Research site, Chicago, Illinois
  - Research site, Maywood, Illinois
  - Research site, Boston, Massachusetts
  - Research site, Detroit, Michigan
  - Research site, Rochester, Minnesota
  - Research site, Omaha, Nebraska
  - Research site, Buffalo, New York
  - Research site, New York, New York
  - Research site, Rochester, New York
  - Research site, Durham, North Carolina
  - Research site, Philadelphia, Pennsylvania
  - Research site, Columbia, South Carolina
  - Research site, Houston, Texas
  - Research site, Charlottesville, Virginia

REFERENCES:
- [Background] Leonard JP, Friedberg JW, Younes A, Fisher D, Gordon LI, Moore J, Czuczman M, Miller T, Stiff P, Cheson BD, Forero-Torres A, Chieffo N, McKinney B, Finucane D, Molina A. A phase I/II study of galiximab (an anti-CD80 monoclonal antibody) in combination with rituximab for relapsed or refractory, follicular lymphoma. Ann Oncol. 2007 Jul;18(7):1216-23. doi: 10.1093/annonc/mdm114. Epub 2007 Apr 29. PMID 17470451